CLINICAL TRIAL: NCT06944184
Title: In Vivo Antibiotic Elution During Two-Stage Knee Revision: A Microdialysis Study
Brief Title: Antibiotic Elution After Two-stage Knee Revision
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B.Sc., University Hospital, Bonn
Other Study IDs: 2024_B
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Periprosthetic Knee Infection
Keywords: two-stage exchange; infection; arthroplasty; PJI; microdialysis; minimal inhibitory concentration; bone cement; treatment monitoring
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients presenting with an infected knee prosthesis
  Interventions: Device: Intraarticular microdialysis

INTERVENTIONS:
Device: Intraarticular microdialysis — The intervention decive is placed during the routine surgery to remove the infected knee prosthesis and implantation of the static cement spacer. A microdialysis catheter is implemented to generate continious intra-articular samples of the knee joint. To ensure complete removal and no damage of the membrane it is inserted via a regular drainage tube. The catheter membrane is placed intra-articularly next to the spacer and continious to an outlet tube for sample collection.

SUMMARY:
The goal of this observational study is to monitor the eluted antibiotic concentrations of gentamicin and vancomycin by a static knee cement spacer in patients being treated for periprosthetic infections of the knee. The main question aims to answer if eluted antibiotics are in a therapeutic range for treatment at sight of infection. Secondarily, local antibiotic concentrations are compared with systemic blood levels, as are systemically applied antibiotics compared to intra-articular concentrations. Intra-articular samples are collected over a 72 hour postoperative period.

DETAILED DESCRIPTION:
The present study moinitors antibiotic concentrations eluted by a static cement knee spacer as two-stage revision treatment of a knee PJI. The static cement spacer consists of COPAL G+V cement containing 2g of vancomycin and 0.5g of gentamicin. Microdialysis is used as a technique for continuous extra cellular sample collection directly from the knee joint cavity. It is implemented guided by a drainage tube during the surgery to remove the infected prosthesis and implement the spacer. Over a 72 hour period samples directly from the knee joint are generated continiously. These are analyzed for the eluded antibiotic concentrations of gentamicin and vancomycin from the knee spacer. Once every 24 hours venous blood samples were collected as well and analyzed for gentamicin and vancomycin and also systemically applied antibiotics (a.e. cefuroxim, clindamycin).

ELIGIBILITY:
Inclusion Criteria:

* clinical indication for a two-staged revision of a knee PJI
* approval for surgery by the orthopedic and anesthesiologic departments
* being over 18 years of age
* written, informed consent after detailed patient information about the study protocol and possible study-dependent risks

Exclusion Criteria:

* known allergies to the antibiotics gentamicin and vancomycin contained in the spacer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ten patients over 18 years with a periprosthetic knee infection after total knee arthorplasty and indication for prosthesis explanation and temporary spacer implantation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
antibiotic concentrations in intra-articular samples | Concentrations are measured for 72 hours after spacer implantation.
  Both locally through the spacer eluted antibiotics (gentamicin and vancomycin) and systemically administered antibiotics (e.g. cefuroxim, clindamycin) are measured in intra-articular knee samples.

SECONDARY OUTCOMES:
Antibiotic concentrations in blood samples | Antibiotic concentrations are measured once every 24 hours after spacer implantation. In total at three time points during the 72 hour observation period.
  Antibiotic concentrations eluted by the spacer (gentamicin, vancomycin) and systemically administered antibiotics (e.g. cefuroxim, clindamycin) are measured in venous blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lazic I, Scheele C, Pohlig F, von Eisenhart-Rothe R, Suren C. Treatment options in PJI - is two-stage still gold standard? J Orthop. 2021 Jan 20;23:180-184. doi: 10.1016/j.jor.2020.12.021. eCollection 2021 Jan-Feb. PMID 33551610
- [Background] Dhanani JA, Parker SL, Lipman J, Wallis SC, Cohen J, Fraser J, Barnett A, Chew M, Roberts JA. Recovery rates of combination antibiotic therapy using in vitro microdialysis simulating in vivo conditions. J Pharm Anal. 2018 Dec;8(6):407-412. doi: 10.1016/j.jpha.2018.07.003. Epub 2018 Jul 6. PMID 30595948
- [Background] Moojen DJ, Hentenaar B, Charles Vogely H, Verbout AJ, Castelein RM, Dhert WJ. In vitro release of antibiotics from commercial PMMA beads and articulating hip spacers. J Arthroplasty. 2008 Dec;23(8):1152-6. doi: 10.1016/j.arth.2007.08.020. Epub 2008 Mar 4. PMID 18534493